CLINICAL TRIAL: NCT01560182
Title: A Phase I/II Clinical Trial of Hematopoietic Stem Cell Gene Therapy for the Treatment of Metachromatic Leukodystrophy
Brief Title: Gene Therapy for Metachromatic Leukodystrophy (MLD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orchard Therapeutics (Industry)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201222; Eudract 2009-017349-77 (Other: IRCCS San Raffaele)
Record Dates: First submitted 2012-03-16; First posted 2012-03-22 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lysosomal Storage Disease; Metachromatic Leukodystrophy
Keywords: OTL-200; Metachromatic Leukodystrophy; Gene Therapy; MLD; Previously GSK2696274
MeSH Terms: conditions — Lysosomal Storage Diseases; Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OTL-200 Gene Therapy (Experimental): CD34+ cells transduced ex vivo with lentiviral vector encoding ARSA cDNA
  Interventions: Genetic: OTL-200 Gene Therapy

INTERVENTIONS:
Genetic: OTL-200 Gene Therapy — Autologous hematopoietic stem/progenitor cells collected from the bone marrow and transduced ex vivo with a Lentiviral vector encoding the human ARSA cDNA
  Other Names: Previously GSK2696274

SUMMARY:
This Phase I/II clinical trial consists of the application of lentiviral vector-based gene therapy to patients affected by Metachromatic Leukodystrophy (MLD), a rare inherited Lysosomal Storage Disorder (LSD) resulting from mutations in the gene encoding the Arylsulfatase A (ARSA) enzyme. The medicinal product consists of autologous CD34+ hematopoietic stem/progenitor cells in which a functional ARSA cDNA is introduced by means of 3rd generation VSV-G pseudotyped lentiviral vectors.

ELIGIBILITY:
Inclusion Criteria:

* Pre-symptomatic MLD patients with the late infantile variant;
* Pre- or early-symptomatic MLD patients with the early juvenile variant;
* Patients for whom parental/guardian signed informed consent has been obtained.

Exclusion Criteria:

* HIV RNA and/or HCV RNA and/or HBV DNA positive patients;
* Patients affected by neoplastic diseases;
* Patients with cytogenetic alterations typical of MDS/AML;
* Patients with end-organ functions or any other severe disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
* Patients enrolled in other trials/other therapeutic approaches that might become available;
* Patient who underwent allogeneic hematopoietic stem cell transplantation in the previous six months;
* Patient who underwent allogenic hematopoietic stem cell transplantation with evidence of residual cells of donor origin.

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-04-09 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Improvement of Gross Motor Function Measure (GMFM) score | 24 months after treatment
  An improvement of 10% of the total GMFM score in treated patients, when compared to the GMFM scores in the historical control MLD population, evaluated 24 months after treatment.
Increase of residual Arylsulfatase A (ARSA) activity | 24 months after treatment
  A significant increase of residual ARSA activity as compared to pre- treatment values, measured in total Peripheral Blood Mononuclear Cells (PBMCs)
Conditioning regimen-related safety | at +60 days after transplantation
  The absence of engraftment failure or delayed hematopoietic reconstitution (prolonged aplasia), defined as Absolute Neutrophil Count (ANC)<500/µl, with no evidence of Bone Marrow (BM) recovery, requiring cellular back-up administration.
Conditioning regimen-related toxicity | 3 years after treatment
  The absence of regimen related toxicity, as determined by a surveillance of adverse events (AEs) (NCI ≥2) and laboratory parameters (NCI ≥3) that will be applied in the short- and long-term follow-up of the treated patients in order to assess the degree of morbidity associated to the conditioning regimen
The short-term safety and tolerability of lentiviral-transduced cell infusion | 48 hours after treatment infusion
  It will be evaluated on the basis of AEs reporting and monitoring of the systemic reactions to cell infusion (fever, tachycardia, nausea and vomiting, joint pain, skin rash). Evaluation will also consist of the absence of Serious Adverse Reactions (SARs) within 48 hours after infusion.
The long-term safety of lentiviral-transduced cell infusion | baseline, 1, 3, 6, and 12 months after treatment, then once a year
  Absence of Replication Competent Lentivirus: Assessed via enzyme-linked immunosorbent assay (ELISA) test for serum human immunodeficiency virus (HIV) p24 antigen. Positive HIV p24 test result is subject to second level testing including: a) DNA PCR for vesicular stomatitis virus G (VSV-G) envelope (PBMC) and b) reverse transcription (RT) PCR for HIV-pol ribonucleic acid (RNA) (plasma).
The long-term safety of lentiviral-transduced cell infusion | baseline, 3, 6 and 12 months after treatment, then once a year
  Absence of Abnormal Clonal Proliferation: monitored by clinical and laboratory surveillance, TCR Vβ repertoire analysis, and bone marrow examination.
The long-term safety of lentiviral-transduced cell infusion | 6 and 12 months after treatment, then once a year
  Lentiviral vector integration site analysis will also be performed

SECONDARY OUTCOMES:
The absence of immune responses against the transgene (immunoblot analyses). | baseline, 3, 6, and 12 months after treatment, then once a year
  Even if immune responses against the functional ARSA enzyme are not expected, treated subjects will be monitored for anti-ARSA antibodies on a defined schedule.
Nerve Conduction Velocity (NCV) Index for Electroneurography (ENG) and total brain MRI score. | 24 months after treatment
  The NCV Index and the total brain MRI score will be compared to scores observed in the historical control MLD population.
  Gross Motor Function Classification for MLD (GMFC-MLD) levels at different ages compared to the historical control MLD population.
Transduced cell engraftment | 12 months after treatment
  Transduced cell engraftment above 4% in bone marrow-derived clonogenic progenitor cells, assessed as the percentage of LV-positive colonies. Vector copy number (VCN) per cell in total PBMC, total BM, and peripheral blood (PB) and bone marrow (BM) cell subpopulations will also be evaluated.
IQ measurement above 55 | 24, 30 and 36 months after treatment
  The measurement of an IQ above 55 (threshold for severe cognitive impairment) at neuro-psychological testings

CONTACTS AND LOCATIONS:
Overall Officials: Orchard Clinical Trials, Study Director — Orchard Therapeutics
Locations (1):
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy

REFERENCES:
- [Background] Biffi A, Capotondo A, Fasano S, del Carro U, Marchesini S, Azuma H, Malaguti MC, Amadio S, Brambilla R, Grompe M, Bordignon C, Quattrini A, Naldini L. Gene therapy of metachromatic leukodystrophy reverses neurological damage and deficits in mice. J Clin Invest. 2006 Nov;116(11):3070-82. doi: 10.1172/JCI28873. PMID 17080200
- [Background] Biffi A, Cesani M, Fumagalli F, Del Carro U, Baldoli C, Canale S, Gerevini S, Amadio S, Falautano M, Rovelli A, Comi G, Roncarolo MG, Sessa M. Metachromatic leukodystrophy - mutation analysis provides further evidence of genotype-phenotype correlation. Clin Genet. 2008 Oct;74(4):349-57. doi: 10.1111/j.1399-0004.2008.01058.x. Epub 2008 Sep 11. PMID 18786133
- [Background] Biffi A, Montini E, Lorioli L, Cesani M, Fumagalli F, Plati T, Baldoli C, Martino S, Calabria A, Canale S, Benedicenti F, Vallanti G, Biasco L, Leo S, Kabbara N, Zanetti G, Rizzo WB, Mehta NA, Cicalese MP, Casiraghi M, Boelens JJ, Del Carro U, Dow DJ, Schmidt M, Assanelli A, Neduva V, Di Serio C, Stupka E, Gardner J, von Kalle C, Bordignon C, Ciceri F, Rovelli A, Roncarolo MG, Aiuti A, Sessa M, Naldini L. Lentiviral hematopoietic stem cell gene therapy benefits metachromatic leukodystrophy. Science. 2013 Aug 23;341(6148):1233158. doi: 10.1126/science.1233158. Epub 2013 Jul 11. PMID 23845948
- [Background] Biffi A, De Palma M, Quattrini A, Del Carro U, Amadio S, Visigalli I, Sessa M, Fasano S, Brambilla R, Marchesini S, Bordignon C, Naldini L. Correction of metachromatic leukodystrophy in the mouse model by transplantation of genetically modified hematopoietic stem cells. J Clin Invest. 2004 Apr;113(8):1118-29. doi: 10.1172/JCI19205. PMID 15085191
- [Background] Capotondo A, Cesani M, Pepe S, Fasano S, Gregori S, Tononi L, Venneri MA, Brambilla R, Quattrini A, Ballabio A, Cosma MP, Naldini L, Biffi A. Safety of arylsulfatase A overexpression for gene therapy of metachromatic leukodystrophy. Hum Gene Ther. 2007 Sep;18(9):821-36. doi: 10.1089/hum.2007.048. PMID 17845130
- [Background] Cesani M, Capotondo A, Plati T, Sergi LS, Fumagalli F, Roncarolo MG, Naldini L, Comi G, Sessa M, Biffi A. Characterization of new arylsulfatase A gene mutations reinforces genotype-phenotype correlation in metachromatic leukodystrophy. Hum Mutat. 2009 Oct;30(10):E936-45. doi: 10.1002/humu.21093. PMID 19606494
- [Derived] Fumagalli F, Calbi V, Gallo V, Zambon AA, Recupero S, Ciotti F, Sarzana M, Fraschini M, Scarparo S, De Mattia F, Miglietta S, Pierini C, Soncini M, Morena F, Montini E, Barzaghi F, Consiglieri G, Ferrua F, Migliavacca M, Tucci F, Fratini ES, Ippolito A, Silvani P, Calvi MR, Clerici A, Corti A, Facchini M, Locatelli S, Sangalli M, Zancan S, Miotto F, Natali Sora MG, Baldoli C, Martino S, Cordoba-Claros A, Moro SL, Gollop ND, Abate J, Yarzi MN, Nutkins P, Shenker A, Calissano M, Brooks J, Richardson A, Campbell L, Filippi M, Naldini L, Cicalese MP, Ciceri F, Bernardo ME, Aiuti A. Long-Term Effects of Atidarsagene Autotemcel for Metachromatic Leukodystrophy. N Engl J Med. 2025 Apr 24;392(16):1609-1620. doi: 10.1056/NEJMoa2405727. PMID 40267426
- [Derived] Fumagalli F, Calbi V, Natali Sora MG, Sessa M, Baldoli C, Rancoita PMV, Ciotti F, Sarzana M, Fraschini M, Zambon AA, Acquati S, Redaelli D, Attanasio V, Miglietta S, De Mattia F, Barzaghi F, Ferrua F, Migliavacca M, Tucci F, Gallo V, Del Carro U, Canale S, Spiga I, Lorioli L, Recupero S, Fratini ES, Morena F, Silvani P, Calvi MR, Facchini M, Locatelli S, Corti A, Zancan S, Antonioli G, Farinelli G, Gabaldo M, Garcia-Segovia J, Schwab LC, Downey GF, Filippi M, Cicalese MP, Martino S, Di Serio C, Ciceri F, Bernardo ME, Naldini L, Biffi A, Aiuti A. Lentiviral haematopoietic stem-cell gene therapy for early-onset metachromatic leukodystrophy: long-term results from a non-randomised, open-label, phase 1/2 trial and expanded access. Lancet. 2022 Jan 22;399(10322):372-383. doi: 10.1016/S0140-6736(21)02017-1. PMID 35065785
- [Derived] Sessa M, Lorioli L, Fumagalli F, Acquati S, Redaelli D, Baldoli C, Canale S, Lopez ID, Morena F, Calabria A, Fiori R, Silvani P, Rancoita PM, Gabaldo M, Benedicenti F, Antonioli G, Assanelli A, Cicalese MP, Del Carro U, Sora MG, Martino S, Quattrini A, Montini E, Di Serio C, Ciceri F, Roncarolo MG, Aiuti A, Naldini L, Biffi A. Lentiviral haemopoietic stem-cell gene therapy in early-onset metachromatic leukodystrophy: an ad-hoc analysis of a non-randomised, open-label, phase 1/2 trial. Lancet. 2016 Jul 30;388(10043):476-87. doi: 10.1016/S0140-6736(16)30374-9. Epub 2016 Jun 8. PMID 27289174